CLINICAL TRIAL: NCT04129554
Title: A Randomized, Double Blind, Placebo-controlled Phase 2b Study to Evaluate Efficacy, Pharmacokinetics, and Safety of 48-week Study Intervention With JNJ 73763989+JNJ 56136379+Nucleos(t)Ide Analog (NA) Regimen Compared to NA Alone in e Antigen Negative Virologically Suppressed Participants With Chronic Hepatitis B Virus Infection
Brief Title: A Study of JNJ 73763989+JNJ 56136379+Nucleos(t)Ide Analog (NA) Regimen Compared to NA Alone in e Antigen Negative Virologically Suppressed Participants With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108679; 73763989PAHPB2002 (Other: Janssen Sciences Ireland UC); 2019-002674-31 (EudraCT Number); NCT04288310 (obsolete NCT alias)
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — JNJ-56136379; entecavir; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- JNJ-73763989+ JNJ-56136379+ NA (Experimental): Participants will receive fixed dose of JNJ-73763989 subcutaneous injection once every 4 weeks along with fixed dose of JNJ-56136379 tablet once daily and nucleos(t)ide analog (NA) treatment (either entecavir [ETV], tenofovir disoproxil fumarate [TDF], or tenofovir alafenamide [TAF]) once daily up to 48 weeks.
  Interventions: Drug: JNJ-73763989; Drug: JNJ-56136379; Drug: Entecavir (ETV) monohydrate; Drug: Tenofovir disoproxil fumarate (TDF); Drug: Tenofovir alafenamide (TAF)
- Placebo for JNJ-73763989+ Placebo for JNJ-56136379+ NA (Placebo Comparator): Participants will receive matching placebo for JNJ-73763989 subcutaneous injection once every 4 weeks with matching placebo for JNJ-56136379 once daily and NA treatment (either ETV, TDF or TAF) once daily up to 48 weeks.
  Interventions: Drug: Placebo for JNJ-73763989; Drug: Placebo for JNJ-56136379; Drug: Entecavir (ETV) monohydrate; Drug: Tenofovir disoproxil fumarate (TDF); Drug: Tenofovir alafenamide (TAF)

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 injection will be administered subcutaneously once every 4 weeks up to 48 weeks.
  Arms: JNJ-73763989+ JNJ-56136379+ NA
Drug: JNJ-56136379 — JNJ-56136379 tablets will be administered orally once daily up to 48 weeks.
  Arms: JNJ-73763989+ JNJ-56136379+ NA
Drug: Placebo for JNJ-73763989 — Matching placebo for JNJ-73763989 will be administered as subcutaneous injection up to 48 weeks.
  Arms: Placebo for JNJ-73763989+ Placebo for JNJ-56136379+ NA
Drug: Placebo for JNJ-56136379 — Matching placebo for JNJ-56136379 tablets will be administered orally up to 48 weeks.
  Arms: Placebo for JNJ-73763989+ Placebo for JNJ-56136379+ NA
Drug: Entecavir (ETV) monohydrate — ETV tablet will be administered orally once daily up to 48 weeks as NA treatment.
Drug: Tenofovir disoproxil fumarate (TDF) — TDF will be administered orally once daily up to 48 weeks as NA treatment.
Drug: Tenofovir alafenamide (TAF) — TAF will be administered orally once daily up to 48 weeks as NA treatment.

SUMMARY:
The purpose of this study is to evaluate the efficacy of 48-week study intervention with JNJ-73763989+JNJ-56136379+nucleos(t)ide analog (NA) regimen compared to NA alone assessed by HBsAg levels. This study is part of HepB Wings Platform Trial (PLATFORMPAHPB2001).

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) is a small deoxyribonucleic acid (DNA) virus that infects the liver and can cause either acute or chronic infection. It consists of a so-called nucleocapsid in which viral DNA is packed with hepatitis B core protein (HBc) and membranous envelope containing hepatitis B surface antigen (HBsAg). Chronic HBV infection may lead to serious illnesses like cirrhosis and hepatocellular carcinoma (HCC). Oral treatment with NAs is effective at suppressing viral DNA formation and lowering virus concentration in blood to levels below lower limit of quantification (LLOQ). JNJ-73763989 is a liver-targeted antiviral therapeutic for subcutaneous injection designed to treat chronic HBV infection via ribonucleic acid interference mechanism but rarely lead to functional cure defined as sustained loss of HBs Ag and HBV DNA in serum. JNJ-56136379 is an orally administered capsid assembly modulator that is being developed for treatment of chronic HBV infection. The aim of study is to evaluate efficacy of 48-week study intervention with JNJ-3989+JNJ-6379+NA regimen compared to NA alone, assessed by HBsAg seroclearance at Week 72 (i.e., 24 weeks after completion of all study interventions at Week 48) without restarting NA treatment in HBeAg negative virologically suppressed chronic hepatitis B (CHB) infected participants who received NA treatment for at least 2 years prior to screening. The study will be 2.3 years and will be conducted in 3 phases: a screening phase (4 weeks), a study intervention phase (48 weeks), and a follow-up phase (48 weeks). Safety will be evaluated by AEs including AEs of special interest to any of the study interventions, clinical laboratory tests, ECGs, vital signs, and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable based on physical examination, medical history, vital signs, electrocardiogram (ECG) at screening
* Chronic hepatitis B virus (HBV) infection with documentation at least 6 months prior to screening
* Hepatitis B e (antigen) (HBeAg)-negative on stable nucleotide analogue (NA) treatment for at least 24 months prior to screening
* Hepatitis B surface antigen (HBsAg) greater than (>) 100 International Units per Milliliter (IU/mL) at screening
* Body mass index (BMI) between 18.0 and 35 kilogram per meter square (kg/m^2), extremes included
* Highly effective contraceptive measures in place for female participants of childbearing potential or male participants with female partners of childbearing potential
* Liver fibrosis stage 0-2 (Metavir) or Fibroscan less than (<) 9 Kilopascal (kPa) at screening

Exclusion Criteria:

* Evidence of infection with hepatitis A, C, D or E virus infection or evidence of human immunodeficiency, virus type 1 (HIV-1) or HIV-2 infection at screening
* History or evidence of clinical signs/symptoms of hepatic decompensation including but not limited to: portal hypertension, ascites, hepatic encephalopathy, esophageal varices or any laboratory abnormalities indicating a reduced liver function as defined in the protocol
* Evidence of liver disease of non-HBV etiology
* History or signs of cirrhosis or portal hypertension (nodules, no smooth liver contour, no normal portal vein, spleen size ≥12 cm) or signs of hepatocellular carcinoma (HCC)
* Significant laboratory abnormalities as defined in the protocol at screening
* Participants with a history of malignancy within 5 years before screening
* Abnormal sinus rhythm or ECG parameters at screening as defined in the protocol
* History of or current cardiac arrhythmia or history or clinical evidence of significant or unstable cardiac disease
* Participants with any current or previous illness for which, in the opinion of the investigator and/or sponsor, participation would not be in the best interest of the participant
* History of or current clinically significant skin disease or drug rash
* Known allergies, hypersensitivity, or intolerance to JNJ-73763989 and JNJ-56136379 or their excipients or to placebo content
* Contraindications to the use of entecavir (ETV), tenofovir disoproxil fumarate (TDF), or tenofovir alafenamide (TAF) per local prescribing information
* Participants who have taken any therapies disallowed per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (41):
- Belgium (5):
  - Cliniques Universitaires Saint Luc, Brussels
  - SGS Belgium NV, Edegem
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- France (7):
  - Hopital Beaujon, Clichy
  - Hopital de La Croix Rousse, Lyon
  - Hopital Saint Joseph, Marseille
  - Hopital Cochin, Paris
  - Chu Rennes Hopital Pontchaillou, Rennes
  - CHU Nancy Brabois, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
- Germany (8):
  - Universitatsklinikum Essen, Essen
  - Universitätsklinikum Johann Wolfgang Goethe- Universität Frankfurt Medizinische Klinik 1, Frankfurt
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - ICH Study Center GmbH & Co. KG, Hamburg
  - University Medical Center, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
- Italy (5):
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Irccs Ospedale Maggiore Di Milano, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Ospedale di Baggiovara, Modena
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Universita degli Studi di Roma 'La Sapienza' - Umberto I Policlinico di Roma, Rome
- Poland (4):
  - Wojewodzki Szpital Obserwacyjno-Zakazny im. Tadeusza Browicza w Bydgoszczy, Bydgoszcz
  - Neutrum Lekarze M.Hlebowicz i Partnerzy spolka partnerska, Gdansk
  - ID Clinic, Mysłowice
  - SP ZOZ Wroclawskie Centrum Zdrowia, Wroclaw
- Spain (6):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Gral. Univ. Valencia, Valencia
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - North Manchester General Hospital, Crumpsall
  - Glasgow Royal Infirmary, Glasgow
  - Grahame Hayton Unit, London
  - Kings College Hospital, London
  - St Georges University of London and St George's University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Agarwal K, Buti M, van Bommel F, Lampertico P, Janczewska E, Bourliere M, Vanwolleghem T, Lenz O, Verbinnen T, Kakuda TN, Mayer C, Jezorwski J, Muenz D, Beumont M, Kalmeijer R, Biermer M, Lonjon-Domanec I. JNJ-73763989 and bersacapavir treatment in nucleos(t)ide analogue-suppressed patients with chronic hepatitis B: REEF-2. J Hepatol. 2024 Sep;81(3):404-414. doi: 10.1016/j.jhep.2024.03.046. Epub 2024 Apr 5. PMID 38583491

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA: Participants received JNJ-73763989 200 mg subcutaneous (SC) injection, once every 4 weeks (q4w), along with JNJ-56136379 250 mg tablet once daily (qd) and NA treatment orally (either entecavir [ETV], tenofovir disoproxil fumarate [TDF] or tenofovir alafenamide [TAF]) qd up to 48 weeks.
- Arm 2: Nucleos(t)Ide Analog (NA): Participants received matching placebo for JNJ-73763989 by SC injection q4w, along with matching placebo for JNJ-56136379 qd and NA treatment orally (either ETV, TDF or TAF) qd up to 48 weeks.
Period: Overall Study
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Started | 85 | 45
Completed | 81 | 40
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA) | Total
Number analyzed (Participants) | 85 | 45 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (10.1) | 47.4 (10.55) | 46 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 16 | 43
  Male | 58 | 29 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 3 | 18
  Not Hispanic or Latino | 66 | 41 | 107
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 8 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 56 | 30 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 7 | 2 | 9
  FRANCE | 14 | 7 | 21
  GERMANY | 7 | 5 | 12
  ITALY | 17 | 5 | 22
  POLAND | 13 | 10 | 23
  SPAIN | 18 | 7 | 25
  UNITED KINGDOM | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Surface Antigen (HBsAg) Seroclearance at Week 72 Without Restarting NA Treatment
Description: Percentage of participants with HBsAg seroclearance at Week 72 (24 weeks after completion of all study interventions at Week 48) without restarting NA treatment was reported. Seroclearance at Week 72 of the treatment defined as a confirmed loss of HBsAg at Week 72. Loss is defined as a baseline HBsAg with a repeat reactive, confirmed or positive result and a post-baseline assessment with a negative result.
Time Frame: Week 72
Population: Modified intent-to-treat (mITT) included all participants who were randomized in the study and received at least one dose of study intervention excluding those participants impacted by the pandemic. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 79 | 39
Percentage of participants | 0.0 | 0.0

2. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant who was administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAE was defined as the AEs occurring after first administration of study intervention (or worsened since then).
Time Frame: From screening up to Week 102
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 85 | 45
Percentage of participants | 85.9 | 80.0

3. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant who was administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAE was defined as the AEs occurring after first administration of study intervention (or worsened since then). SAEs included any untoward medical occurrence that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the off spring of a study participant.
Time Frame: From screening up to 102 weeks
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 85 | 45
Percentage of participants | 3.5 | 8.9

4. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance at Week 48
Description: Percentage of participants with hepatitis B surface antigen (HBsAg) seroclearance at Week 48 was reported. Seroclearance at Week 48 of the treatment defined as a confirmed loss of HBsAg at Week 48. Loss is defined as a baseline HBsAg with a repeat reactive, confirmed or positive result and a post-baseline assessment with a negative result.
Time Frame: Week 48
Population: mITT included all participants who were randomized in the study and received at least one dose of study intervention excluding those participants impacted by the pandemic. Here, 'N' (number of subjects analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 76 | 41
Percentage of participants | 0 | 0

5. Secondary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Less Than (<) Lower Limit of Quantification (LLOQ) at Week 48
Description: Percentage of participants with HBV DNA <LLOQ (20 international units per milliliters [IU/mL]) at Week 48 was reported.
Time Frame: Week 48
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 75 | 41
Percentage of participants | 97.3 | 100

6. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance at Week 96 (48 Weeks After Stopping All Study Interventions at Week 48 Without Restarting NA Treatment)
Description: Percentage of participants with HBsAg seroclearance at Week 96 (48 weeks after stopping all study interventions at Week 48 without restarting NA treatment) was reported. Seroclearance at Week 96 of the treatment defined as a confirmed loss of HBsAg at Week 96. Loss is defined as a baseline HBsAg with a repeat reactive, confirmed or positive result and a post-baseline assessment with a negative result. Missing values were imputed by last observation carried forward (LOCF).
Time Frame: Week 96
Population: mITT included all participants who were randomized in the study and received at least one dose of study intervention excluding those participants impacted by the pandemic.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 84 | 44
Percentage of participants | 0.0 | 0.0

7. Secondary Outcome: Percentage of Participants With (Sustained) Reduction, Suppression, and/or Seroclearance
Description: Percentage of participants with (sustained) reduction, suppression, and/or seroclearance considering single and multiple markers (such as hepatitis B surface antigen [HBsAg] and HBV DNA) (HBsAg >= lower limit of quantification [LLOQ] and HBV DNA<2000 IU/mL; HBsAg >= LLOQ and LLOQ <= HBV DNA < 2000 IU/mL) off-treatment was reported.
Time Frame: Baseline (Day 1) up to Week 96
Population: mITT included all participants, who were randomized in the study and received at least one dose of study intervention excluding those participants impacted by the pandemic. Here, 'N' (number of participants analyzed) included participants with blood marker data.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 71 | 28
Percentage of participants
  HBsAg>=LLOQ and HBVDNA<2000 IU/mL | 23.9 | 3.6
  HBsAg>=LLOQ and LLOQ<=HBV DNA <2000 IU/mL | 64.8 | 64.3

8. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion at Week 96
Description: Percentage of participants with HBsAg seroconversion were reported. HBsAg seroconversion was defined as HBsAg seroclearance together with appearance of anti-hepatitis B surface (HBs) or anti-hepatitis e (HBe) antibodies, respectively.
Time Frame: Week 96
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 81 | 39
Percentage of participants | 0 | 0

9. Secondary Outcome: Change From Baseline in HBsAg Values at Weeks 48, 72, and 96
Description: Change from baseline in HBsAg values was reported.
Time Frame: Baseline (Day 1), Weeks 48, 72, and 96
Population: mITT included all participants who were randomized in the study and received at least one dose of study intervention excluding those participants impacted by the pandemic. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number evaluable) signifies number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 81 | 41
log10 IU/mL
  Week 48: number analyzed (Participants) | 76 | 41
  Week 48 | -1.89 (0.522) | -0.06 (0.082)
  Week 72: number analyzed (Participants) | 79 | 39
  Week 72 | -1.76 (0.658) | -0.25 (0.563)
  Week 96: number analyzed (Participants) | 81 | 40
  Week 96 | -1.46 (0.661) | -0.49 (0.783)

10. Secondary Outcome: Change From Baseline in HBV DNA Values at Weeks 48, 72, and 96
Description: Change from baseline in HBV DNA values was reported. Participants were considered as virologically suppressed if they were on stable HBV treatment (receiving NA treatment [ETV, TDF, or TAF)] for at least 24 months prior to screening and were on the same dose of NA treatment regimen for at least 3 months at the time of screening, and had serum HBV DNA less than (<)60 IU/mL on 2 sequential measurements at least 6 months and had documented alanine aminotransferase values <2.0* upper limit of normal on 2 sequential measurements at least 6 months apart.
Time Frame: Baseline (Day 1), Weeks 48, 72, and 96
Population: mITT included as all participants who were randomized in the study and received at least one dose of study intervention excluding those participants impacted by the pandemic. Here, 'N' (number of participants analyzed) signifies that no participants were available for change from baseline HBV DNA analysis because all participants were virologically suppressed, thereby planned data collection and analysis was not performed and thus, no data was reported for this outcome measure.
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Achieve First HBsAg Seroclearance
Description: Time to achieve first HBsAg seroclearance was defined as the number of days between the date of first study treatment intake and the date of the first occurrence of HBsAg seroclearance.
Time Frame: Baseline (Day 1) up to Week 96
Population: mITT included all participants who were randomized in the study and received at least one dose of study intervention excluding those participants impacted by the pandemic. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 83 | 44
Days | NA [NA to NA] — Here, NA indicates that median and full range for the first occurrence of HBsAg seroclearance after first intake of study treatment was not estimable because of less number of events. | NA [NA to NA] — Here, NA indicates that median and full range for the first occurrence of HBsAg seroclearance after first intake of study treatment was not estimable because of less number of events.

12. Secondary Outcome: Percentage of Participants With Reduction of More Than (>) 1 log10 IU/mL in HBsAg Levels From Baseline
Description: Percentage of participants with reduction of >1 log10 in HBsAg Levels IU/mL from baseline was reported.
Time Frame: Baseline (Day 1) up to Week 96
Population: mITT included as all participants who were randomized in the study and received at least one dose of study intervention excluding those participants impacted by the pandemic. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 81 | 40
Percentage of participants | 81.5 | 12.5

13. Secondary Outcome: Percentage of Participants With HBsAg Levels Less Than (<) 100 IU/mL at Weeks 48, 72, and 96
Description: Percentage of participants with HBsAg Levels <100 IU/mL at Weeks 48, 72, and 96 was reported.
Time Frame: Weeks 48, 72, and 96
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 81 | 41
Percentage of participants
  Week 48: number analyzed (Participants) | 76 | 41
  Week 48 | 71.1 | 2.4
  Week 72: number analyzed (Participants) | 79 | 39
  Week 72 | 67.1 | 10.3
  Week 96: number analyzed (Participants) | 81 | 40
  Week 96 | 46.9 | 15.0

14. Secondary Outcome: Percentage of Participants With HBV DNA Levels Less Than (<) LLOQ From Baseline up to Week 96 (End of Study)
Description: Percentage of Participants with HBV DNA levels <LLOQ (20 IU/mL) was reported.
Time Frame: Baseline (Day 1) up to Week 96
Population: mITT included as all participants who were randomized in the study and received at least one dose of study intervention excluding those participants impacted by the pandemic. Here, 'N' (number of participants analyzed) included participants with blood marker data.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 71 | 28
Percentage of participants | 23.9 | 3.6

15. Secondary Outcome: Percentage of Participants With Flares
Description: Percentage of participants with flares (virologic, biochemical and clinical flares) was reported. Biochemical flare was defined as confirmed alanine transaminase flare and/or aspartate aminotransferase flare >=3*upper limit of normal and >=3*nadir. The start of a confirmed virologic flare was defined as the first date of two consecutive visits with HBV DNA >200 IU/mL. The end date of the same confirmed virologic flare was defined as the first date when HBV DNA value returns to less than or equal to (<=)200 IU/mL or the date of NA treatment restart, whichever comes first. Clinical flare was defined as participants with both virologic and biochemical flare.
Time Frame: Baseline (Day 1) up to Week 96
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 77 | 41
Percentage of participants
  Virologic Flare (HBV DNA > 200 - =<2000 IU/mL): number analyzed (Participants) | 75 | 40
  Virologic Flare (HBV DNA > 200 - =<2000 IU/mL) | 38.7 | 25.0
  Virologic Flare (HBV DNA>2000 - =< 20000 IU/mL): number analyzed (Participants) | 75 | 40
  Virologic Flare (HBV DNA>2000 - =< 20000 IU/mL) | 24.0 | 30.0
  Virologic Flare (HBV DNA >20000 - =<100000 IU/mL): number analyzed (Participants) | 75 | 40
  Virologic Flare (HBV DNA >20000 - =<100000 IU/mL) | 8.0 | 10.0
  Virologic Flare (HBV DNA >100000 IU/mL): number analyzed (Participants) | 75 | 40
  Virologic Flare (HBV DNA >100000 IU/mL) | 2.7 | 27.5
  Alanine Transaminase Flare | 3.9 | 19.5
  Aspartate Aminotransferase Flare | 1.3 | 14.6
  Clinical Flare: HBV DNA > 200 - =<2000IU/mL: number analyzed (Participants) | 75 | 40
  Clinical Flare: HBV DNA > 200 - =<2000IU/mL | 0.0 | 0.0
  Clinical Flare: HBV DNA > 2000 - =<20000IU/mL: number analyzed (Participants) | 75 | 40
  Clinical Flare: HBV DNA > 2000 - =<20000IU/mL | 1.3 | 0.0
  Clinical Flare: HBV DNA > 20000 - =<100000IU/mL: number analyzed (Participants) | 75 | 40
  Clinical Flare: HBV DNA > 20000 - =<100000IU/mL | 1.3 | 0.0
  Clinical Flare: HBV DNA > 100000 IU/mL: number analyzed (Participants) | 75 | 40
  Clinical Flare: HBV DNA > 100000 IU/mL | 1.3 | 27.5

16. Secondary Outcome: Percentage of Participants With Virologic Breakthrough
Description: Percentage of participants with virologic breakthrough defined as confirmed on-treatment HBV DNA increase by more than (>) 1 log10 IU/mL from nadir level or confirmed on treatment level >200 IU/mL in participants who had HBV DNA level below <LLOQ of the HBV DNA assay was reported.
Time Frame: Baseline (Day 1) up to Week 48
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 84 | 44
Percentage of participants | 0.0 | 0.0

17. Secondary Outcome: Percentage of Participants Requiring NA Re-Treatment During Follow-up
Description: Percentage of participants requiring NA re-treatment (either ETV, TDF, or TAF) during follow-up was reported.
Time Frame: Baseline (Day 1) up to Week 96
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 77 | 41
Percentage of participants | 9.1 | 26.8

18. Secondary Outcome: Correlation Coefficient Between On-treatment HBsAg Change From Baseline With On-treatment HBV Blood Markers and Baseline Characteristics
Description: Correlation coefficient between on-treatment HBsAg change from baseline with on-treatment HBV blood markers and baseline characteristics was reported at different timepoints (against age, baseline NA treatment duration, HBsAg value at baseline, HBsAg values at Weeks 24 and 48).
Time Frame: Baseline (Day 1) to Week 96
Population: as for outcome 11
Measure: Number; unit: correlation coefficient
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
Number analyzed (Participants) | 79 | 39
correlation coefficient
  Age | 0.2860 | 0.1746
  Baseline NA treatment duration: number analyzed (Participants) | 78 | 39
  Baseline NA treatment duration | 0.2381 | 0.4324
  HBsAg value at baseline | -0.9970 | -0.5923
  HBsAg at Week 24: number analyzed (Participants) | 74 | 39
  HBsAg at Week 24 | 0.9983 | 0.7120
  HBsAg at Week 48: number analyzed (Participants) | 74 | 39
  HBsAg at Week 48 | 0.9982 | 0.8065

19. Secondary Outcome: Observed Plasma Concentration at Predose (C[Predose]) of JNJ-73763976 (Molecule of JNJ-73763989)
Description: C(predose) was defined as the observed plasma concentration of JNJ-73763976 (a molecule of JNJ-73763989) at predose of JNJ-73763989. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Predose at Weeks 4, 8, 12, and 16
Population: Pharmacokinetic (PK) analysis set included all participants who had received at least 1 dose of any of the study interventions and had at least 1 valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure. NA (nucleos[t]ide analog) was tenofovir disoproxil fumarate (TDF).
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 18
nanogram/milliliter (ng/mL) | NA (NA) — Here, NA indicated that data was below quantification limit (<2.1 ng/mL).

20. Secondary Outcome: Maximum Observed Analyte Concentration (Cmax) of JNJ-73763976 (Molecule of JNJ-73763989)
Description: Cmax was defined as the maximum observed concentration of JNJ-73763976 (molecule of JNJ-73763989). PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: PK analysis set included participants who had received at least 1 dose of any of the study interventions and had at least 1 valid blood sample drawn for PK analysis. NA was TDF. Here, 'N' (number analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 18
ng/mL | 1111 (716) [lower limit 716]

21. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-73763976 (Molecule of JNJ-73763989)
Description: tmax was defined as the time to reach the maximum observed plasma concentration of JNJ-73763976 (molecule of JNJ-73763989). PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: PK analysis set included participants who had received at least 1 dose of any of the study interventions and had at least 1 valid blood sample drawn for PK analysis. Here, 'N' (number of participants analyzed) signifies participants who were evaluable for this outcome measure. NA was TDF.
Measure: Median (Full Range); unit: Hour
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 18
Hour | 6.00 (1.00) [1.00 to 10.00]

22. Secondary Outcome: Observed Plasma Concentration at 24 Hour Postdose (C[24h]) of JNJ-73763976 (Molecule of JNJ-73763989)
Description: C(24h) was defined as the observed plasma concentration of JNJ-73763976 (a molecule of JNJ-73763989) at 24 h postdose of JNJ-73763989. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: 24 hours postdose at Weeks 4, 8, 12, and 16
Population: PK analysis set included participants who had received at least 1 dose of any of the study interventions and had at least 1 valid blood sample drawn for PK analysis. Here, 'N' (number analyzed) signifies number of participants analyzed for this outcome measure. NA was TDF.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 18
ng/mL | 275 (161) [lower limit 161]

23. Secondary Outcome: Area Under the Analyte Concentration Versus Time Curve From Time 0 to 24 Hours (AUC[0-24h]) of JNJ-73763976 (Molecule of JNJ-73763989)
Description: AUC(0-24h) was defined as the area under the concentration of JNJ-73763976 (a molecule of JNJ-73763989) versus time curve from time 0 to 24 hours of JNJ-73763989. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: 0 to 24 hours postdose at Weeks 4, 8, 12, and 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*h/mL)
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 17
nanogram*hour/milliliter (ng*h/mL) | 17833 (9670) [lower limit 9670]

24. Secondary Outcome: Maximum Observed Analyte Concentration (Cmax) of JNJ-73763976 (Molecule of JNJ-73763989) Dose Normalized to 1 mg (Cmax[Dose Normalized])
Description: Cmax(Dose Normalized) was defined as the maximum observed concentration of JNJ-73763976 (a molecule of JNJ-73763989) dose normalized to 1 mg. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 18
ng/mL/mg | 8.34 (5.37) [lower limit 5.37]

25. Secondary Outcome: Area Under the Analyte Concentration Versus Time Curve From Time 0 to 24 Hours of JNJ-73763976 (Molecule of JNJ-73763989) Dose Normalized to 1 mg (AUC[0-24h], Dose Normalized)
Description: AUC([0-24h], Dose Normalized) was defined as the area under the concentration of JNJ-73763976 (molecule of JNJ-73763989) versus time curve from time 0 to 24 hours of JNJ-73763989 dose normalized to 1 mg. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: 0 to 24 hours post-dose at Weeks 4, 8, 12, and 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng*h/mL/mg
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 17
ng*h/mL/mg | 134 (72.5) [lower limit 72.5]

26. Secondary Outcome: Observed Plasma Concentration at Predose (C[Predose]) of JNJ-73763924 (Molecule of JNJ-73763989)
Description: C(predose) was defined as the observed plasma concentration of JNJ-73763924 (a molecule of JNJ-73763989) at predose of JNJ-73763989. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Predose at Weeks 4, 8, 12, and 16
Population: PK analysis set was defined as participants who had received at least 1 dose of any of the study interventions and had at least 1 valid blood sample drawn for PK analysis. Here, 'N' (number analyzed) signifies number of participants analyzed at each specified outcome measure. NA was TDF.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 18
ng/mL | NA (NA) — Here, NA indicates that mean and standard deviation could not be estimated as data was below quantification limit (<2.1 ng/mL).

27. Secondary Outcome: Maximum Observed Analyte Concentration (Cmax) of JNJ-73763924 (Molecule of JNJ-73763989)
Description: Cmax was defined as the maximum concentration of JNJ-73763924 (molecule of JNJ-73763989). PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 18
ng/mL | 222 (142) [lower limit 142]

28. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-73763924 (Molecule of JNJ-73763989)
Description: tmax was defined as the time to reach the maximum observed plasma concentration of JNJ-73763924 (molecule of JNJ-73763989). PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 22
Measure: Median (Full Range); unit: Hour
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 18
Hour | 5.07 (1.00) [1.00 to 8.03]

29. Secondary Outcome: Observed Plasma Concentration at 24 Hour Postdose (C[24h]) of JNJ-73763924 (Molecule of JNJ-73763989)
Description: C(24h) was defined as the observed plasma concentration of JNJ-73763924 (molecule of JNJ-73763989) at 24 h postdose of JNJ-73763989. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: 24 hours postdose at Weeks 4, 8, 12, and 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 17
ng/mL | 35.0 (25.5) [lower limit 25.5]

30. Secondary Outcome: Area Under the Analyte Concentration Versus Time Curve From Time 0 to 24 Hour (AUC[0-24h]) of JNJ-73763924 (Molecule of JNJ-73763989)
Description: AUC(0-24h) was defined as the area under the concentration of JNJ-73763924 (molecule of JNJ-73763989) versus time curve from time 0 to 24 hour of JNJ-73763989. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: 0 to 24 hours postdose at Weeks 4, 8, 12, and 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 17
ng*h/mL | 3386 (1930) [lower limit 1930]

31. Secondary Outcome: Maximum Observed Analyte Concentration (Cmax) of JNJ-73763924 (Molecule of JNJ-73763989) Dose Normalized to 1 mg (Cmax[Dose Normalized])
Description: Cmax(Dose Normalized) was defined as the maximum observed analyte concentration of JNJ-73763924 (molecule of JNJ-73763989) dose normalized to 1 mg. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: nanogram/milliliter/milligram (ng/mL/mg)
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 18
nanogram/milliliter/milligram (ng/mL/mg) | 3.33 (2.14) [lower limit 2.14]

32. Secondary Outcome: Area Under the Analyte Concentration Versus Time Curve From Time 0 to 24 Hours of JNJ-73763924 (Molecule of JNJ-73763989) Dose Normalized to 1 mg (AUC[0-24h], Dose Normalized)
Description: AUC([0-24h], Dose Normalized) was defined as the area under the analyte concentration JNJ-73763924 (a molecule of JNJ-73763989) versus time curve from time 0 to 24 hours of JNJ-73763989 dose normalized to 1 mg. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: 0 to 24 hours postdose at Weeks 4, 8, 12, and 16
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng*h/mL/mg
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 17
ng*h/mL/mg | 50.8 (28.9) [lower limit 28.9]

33. Secondary Outcome: Observed Plasma Concentration at Predose (C[Predose]) of JNJ-56136379
Description: C(predose) was defined as the observed plasma concentration at predose of JNJ-56136379. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Predose at Weeks 4, 8, 12, and 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 12
ng/mL | 10812 (2430) [lower limit 2430]

34. Secondary Outcome: Maximum Observed Analyte Concentration (Cmax) of JNJ-56136379
Description: Cmax was defined as the maximum observed concentration of JNJ-56136379. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 12
ng/mL | 14754 (4318) [lower limit 4318]

35. Secondary Outcome: Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-56136379
Description: tmax was defined as the time to reach the maximum observed plasma concentration of JNJ-56136379. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 22
Measure: Median (Full Range); unit: Hour
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 12
Hour | 4.00 (0.0) [0.0 to 24.17]

36. Secondary Outcome: Observed or Predicted Concentration at the End of a Dosing Interval (Ctau) of JNJ-56136379
Description: Ctau was defined as the observed or predicted concentration at the end of a dosing interval of JNJ-56136379. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 11
ng/mL | 12763 (4959) [lower limit 4959]

37. Secondary Outcome: Area Under the Analyte Concentration Versus Time Curve During a Dosing Interval at Steady State (AUCtau) of JNJ-56136379
Description: AUCtau was defined as the area under the analyte concentration versus time curve during a dosing interval at steady state of JNJ-56136379. PK sample collection was done based on the availability of the participants at Weeks 4, 8, 12, or 16 and thus collected data were averaged and reported in this outcome measure.
Time Frame: Weeks 4, 8, 12, and 16: at Predose, 15 minutes, 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: PK analysis set included participants who have received at least 1 dose of any of the study interventions and have at least 1 valid blood sample drawn for PK analysis. Here, 'N' (number analyzed) signifies number of participants analyzed for this outcome measure. NA was TDF.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA
Number analyzed (Participants) | 12
ng*h/mL | 282458 (79118) [lower limit 79118]

ADVERSE EVENTS:
Time Frame: Up to Week 102 (including 6 weeks of screening)
Description: The safety analysis set included all participants who received at least 1 dose of study drug.
Arm/Group | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA | Arm 2: Nucleos(t)Ide Analog (NA)
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/45
Serious Adverse Events (participants affected / at risk) | 3/85 | 4/45
Other Adverse Events (participants affected / at risk) | 71/85 | 36/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA (N=85) | Arm 2: Nucleos(t)Ide Analog (NA) (N=45)
Vertigo (Ear and labyrinth disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Subacute Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Covid-19 (Infections and infestations) | 1 | 0
Cytomegalovirus Infection Reactivation (Infections and infestations) | 1 | 0
Hepatitis B Reactivation (Infections and infestations) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: JNJ-73763989 (200 Milligrams [mg])+JNJ-56136379 (250 mg)+NA (N=85) | Arm 2: Nucleos(t)Ide Analog (NA) (N=45)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Sinus Arrhythmia (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 2
Ocular Hyperaemia (Eye disorders) | 2 | 0
Visual Impairment (Eye disorders) | 0 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 3 | 0
Dental Caries (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 6
Duodenogastric Reflux (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric Polyps (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 0 | 1
Lip Ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 2
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1
Asthenia (General disorders) | 12 | 4
Chest Discomfort (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 1
Chills (General disorders) | 2 | 0
Fatigue (General disorders) | 11 | 5
Feeling Abnormal (General disorders) | 2 | 0
Illness (General disorders) | 2 | 0
Influenza Like Illness (General disorders) | 3 | 0
Injection Site Haematoma (General disorders) | 0 | 1
Injection Site Pain (General disorders) | 4 | 0
Injection Site Rash (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Pain (General disorders) | 2 | 0
Peripheral Swelling (General disorders) | 1 | 1
Pyrexia (General disorders) | 8 | 3
Suprapubic Pain (General disorders) | 0 | 1
Vaccination Site Pain (General disorders) | 3 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1
Seasonal Allergy (Immune system disorders) | 3 | 0
Bronchitis (Infections and infestations) | 2 | 0
Covid-19 (Infections and infestations) | 17 | 4
Herpes Zoster (Infections and infestations) | 0 | 1
Infected Dermal Cyst (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 10 | 5
Pharyngitis (Infections and infestations) | 2 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 1
Rhinitis (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 2 | 0
Tooth Abscess (Infections and infestations) | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 0
Viral Infection (Infections and infestations) | 0 | 1
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 6 | 11
Amylase Increased (Investigations) | 1 | 2
Aspartate Aminotransferase Increased (Investigations) | 3 | 4
Blood Bilirubin Increased (Investigations) | 3 | 0
Blood Iron Decreased (Investigations) | 0 | 1
Blood Phosphorus Decreased (Investigations) | 0 | 1
Blood Pressure Diastolic Increased (Investigations) | 2 | 0
Creatinine Renal Clearance Decreased (Investigations) | 2 | 0
Crystal Urine Present (Investigations) | 0 | 1
Glomerular Filtration Rate Abnormal (Investigations) | 0 | 1
Glomerular Filtration Rate Decreased (Investigations) | 18 | 4
Hepatitis B Dna Increased (Investigations) | 2 | 3
Lipase Increased (Investigations) | 2 | 2
Sars-Cov-2 Test Positive (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 9 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 19 | 10
Hypoaesthesia (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 2
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 4
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Sleep Disorder (Psychiatric disorders) | 0 | 2
Chromaturia (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 2
Polyuria (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 3 | 0
Semenuria (Renal and urinary disorders) | 0 | 1
Urine Odour Abnormal (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Breast Mass (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 1
Testicular Pain (Reproductive system and breast disorders) | 1 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Haematoma (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 11 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/54/NCT04129554/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT04129554/SAP_001.pdf